CLINICAL TRIAL: NCT03248089
Title: Spanish Lung Liquid vs. Invasive Biopsy Program
Brief Title: Spanish Lung Liquid vs. Invasive Biopsy Program (SLLIP)
Acronym: SLLIP
Status: Completed | Type: Observational
Sponsor: MedSIR (Other)
Collaborators: Guardant Health, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: MedOPP125
Record Dates: First submitted 2017-08-01; First posted 2017-08-14 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Approximately 20 mL of peripheral blood will be collected in StreckTM tubeS. cfDNA will be drawn following blood withdraws following standard of care of the participating site, which would be, before treatment (v2); on the same date as the first standard of care labs (V3), which would be approximately 2 weeks (14 days) into first-line treatment and after one year from enrollment or upon progression whichever occurs first (EoS visit).
  enrollment or upon progression whichever occurs first (EoS visit).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

INTERVENTIONS:
Diagnostic Test: Guardant360 — Cell-free circulating tumor DNA (cfDNA) targeted next-generation sequencing (NGS) panel.

SUMMARY:
Tumor Derived cell free DNA (cfDNA) is increasingly used in the clinic to obtain genotype information about lung cancer, but its concordance with concurrent tumor-derived sequenced data is not known. The primary objective of this study is to demonstrate the non-inferiority of cfDNA-based versus tumor tissue-based genotyping.

DETAILED DESCRIPTION:
Primary objective:

To demonstrate the non-inferiority of cfDNA-based versus tumor tissue-based genotyping as it pertains to the detection of clinically-actionable biomarkers in first line, treatment naïve, metastatic non-squamous NSCLC.

The following secondary objectives will be studied:

* Turn around Time (TAT) of cfDNA vs. tissue results.
* Time to treatment (TtT) initiation.
* Quantity not sufficient rate (QNS) of tissue for clinically-actionable biomarker testing.
* Tumor Not Detected (TND) rate of cfDNA in blood.
* Rescue rate of QNS samples using cfDNA-derived genotyping.
* Rate response for patients that are actionable biomarker positive (either in cDNA or tissue) treated with target-drugs according investigator criteria. Up to three RECIST assessments per patient will be retrospectively done by external personnel (no investigational team).
* Rate of discovery of genomically mediated, acquired resistance to targeted therapies in the biomarker-positive subsets.

ELIGIBILITY:
Inclusion Criteria:

* Patients biopsy-proven, metastatic, previously untreated, non-squamous non-small cell lung cancer (NSCLC). Patients may have received adjuvant cytotoxic chemotherapy, but not targeted neo-adjuvant or adjuvant therapy.
* Age ≥ 18 years
* Ability to understand a written informed consent document, and the willingness to sign it.
* Willingness to provide blood sample at the time points defined in Table 1 [pre-treatment, Day 14 (+/- 7 days) and End of Study].
* Patient has or will have standard-of-care tissue genotyping ordered.
* Stable Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2

Exclusion Criteria:

* Pregnancy, recorded from clinical records
* Any concurrent, non-cutaneous, malignancy (with the exception of early stage non-invasive cervical cancer). Any prior cancer must have occurred more than 5 years prior with no evidence of currently active disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 182 patients with previously untreated non-small cell lung cancer (NSCLC), non-squamous subtype will be recruited for this study, wherein Cell free DNA (cfDNA) will be compared to biopsy-based tumor sequencing
Sampling Method: Probability Sample
Enrollment: 186 (Actual)
Dates: Start 2016-07 (Actual); Primary Completion 2017-07 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Non-inferiority of cell free DNA (cfDNA)-based versus tumor tissue-based genotyping | From date of inclusion until 12 months from enrollment follow-up or upon progression, death or withdrawal from study participation, whichever occurs first.
  Demonstrate the non-inferiority of cell free DNA (cfDNA)-based versus tumor tissue-based genotyping as it pertains to the detection of clinically-actionable biomarkers in first line, treatment naïve, metastatic non-squamous Non-small cell lung cancer (NSCLC).

SECONDARY OUTCOMES:
Turn around Time (TAT) of cell free DNA (cfDNA) vs. tissue results | From pre-treatment visit until month 12 or upon progression, whichever occurs first
  Turn around Time (TAT) of cell free DNA (cfDNA) vs. tissue results
Time to treatment (TtT) initiation | From the date of enrollment in the study until D1 (treatment initiation)
  Time to treatment (TtT) initiation
Quantity not sufficient rate (QNS) of tissue | From day 0 to pre-treatment visit
  Quantity not sufficient rate (QNS) of tissue for clinically-actionable biomarker testing
Tissue Incomplete (TI) rate of tissue | From day 0 to pre-treatment visit
  Tissue Incomplete (TI) rate of tissue for National Cancer Center Network (NCCN) biomarker testing
Tumor Not Detected (TND) rate of cell free DNA (cfDNA) | From pre-treatment visit until month 12 or upon progression, whichever occurs first
  Tumor Not Detected (TND) rate of cell free DNA (cfDNA) in blood
Rescue rate of Quantity not sufficient (QNS) samples using cell free DNA (cfDNA)-derived genotyping | From pre-treatment visit until month 12 or upon progression, whichever occurs first
  Rescue rate of Quantity not sufficient (QNS) samples using cell free DNA (cfDNA)-derived genotyping
Rate response for patients that are actionable biomarker positive (either in cell DNA (cDNA) or tissue) treated with target-drugs | From visit 0 until month 12 or upon progression, whichever occurs first
  Rate response for patients that are actionable biomarker positive (either in cell DNA (cDNA) or tissue) treated with target-drugs according investigator criteria.
Rate of discovery of genomically mediated, acquired resistance to targeted therapies | From visit 0 until month 12 or upon progression, whichever occurs first
  Rate of discovery of genomically mediated, acquired resistance to targeted therapies in the biomarker-positive subsets.

CONTACTS AND LOCATIONS:
Overall Officials: Rafael Rosell, Principal Investigator — IOR
Locations (7):
- Spain (7):
  - H. Can Ruti, Badalona
  - Dexeus, Barcelona
  - H. del Mar, Barcelona
  - H. Sant Pau, Barcelona
  - H. Vall Hebrón, Barcelona
  - ICO Bellvitge, L'Hospitalet de Llobregat
  - H. Arnau de Vilanova, Valencia

IPD SHARING:
Plan to Share IPD: No